CLINICAL TRIAL: NCT04945512
Title: Efficacy of Epidural Analgesia Initiated in the Preoperative Period in Lower Extremity Osteosarcoma
Brief Title: Efficacy of Epidural Analgesia in Lower Extremity Osteosarcoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Nur Canbolat, Principle Invastigator, M.D., Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020/1831
Record Dates: First submitted 2021-06-08; First posted 2021-06-30 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Osteosarcoma; Analgesia
Keywords: epidural analgesia; lower extremity osteosarcoma
MeSH Terms: conditions — Osteosarcoma; Agnosia | interventions — Analgesia, Epidural

STUDY DESIGN:
Intervention Model Description: Study group and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group; Epidural catheter and PCA (Experimental): Epidural catheter will be placed in the preoperative period. After induction, 10 ml of 0.25% bupivacaine will be administered through the epidural catheter and bupivacaine PCA will be started.
  Interventions: Procedure: Epidural Analgesia
- Control group; No block, IC PCA (No Intervention): Postoperative pain control will be achieved with intravenous morphine PCA.

INTERVENTIONS:
Procedure: Epidural Analgesia — In the anesthesia preparation room, an epidutal catheter will be placed with a toue needle through the L4-5 spinal space. After induction of general anesthesia, 10 ml of 0.25% bupivacaine will be injected through the epidural catheter.Afterwards, peroperative and postoperative analgesia will be provided with epidural PCA.
  Arms: Study group; Epidural catheter and PCA

SUMMARY:
In this study, the investigators aim to reduce complications in orthopedic malignancy surgeries and to increase the quality of life of patients who will be operated on.

DETAILED DESCRIPTION:
In the preoperative period, the participants will be taken to the block room. The participants will be monitored, standard sedation will be applied.

Patients in the first group will be provided with preoperative and peroperative analgesia with an epidural catheter. The second group patient will be get no block. Afterwards, both groups will be operated under similar general anesthesia conditions. A patient-controlled analgesia device will be attached to each group of participants and their postoperative follow-up will be made.

ELIGIBILITY:
Inclusion Criteria:

* accepting the study protocol,
* age older than 18 years and younger than 80 years,
* undergoing lower extremity osteosarcoma surgery
* the American Society of Anesthesiologist (ASA) physical status of I-II-III

Exclusion Criteria:

* infection at the injection site
* coagulation disorder
* patients with central nervous system related disease
* septic patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-11-07 (Actual); Primary Completion 2022-08-20 (Estimated); Study Completion 2022-09-20 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | 48 hours
  miligram
Measurement of postoperative pain | 48 hours
  VAS (visual analog scale) (0: no pain, 10: the worst pain imaginable)

SECONDARY OUTCOMES:
Amount of peroperative bleeding | During surgery
  Mililiter
Amount of postoperative bleeding | 48 Hours
  Mililiter
Postoperative complications | postoperative period up to 3 days
  yes/no
Intensive care unit stay | 48 hours
  hours
Hospital stay | 72 hours
  hours
Patient satisfaction | Will be done 3 times 1- a day after surgery 2- in the 1st week follow up after surgery 3- in the 1st month follow-up after surgery
  5-point Likert scale: very satisfied (= 5), satisfied (= 4), neutral (= 3), dissatisfied (= 2) and very dissatisfied (= 1)
Beck Depression Inventory (BDI) | Will be done 2 times 1- on pre-operative hospitalization 2- in the 1st month follow-up after surgery]
  0-9: indicates minimal depression 10-18: indicates mild depression 19-29: indicates moderate depression 30-63: indicates severe depression

CONTACTS AND LOCATIONS:
Overall Officials: Gizem Toydemir, MD, Principal Investigator — Istanbul Unıversity, Istanbul Faculty of Medicine, Anesthesiology
Locations (1):
- Istanbul University, Faculty of Medicine, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rawal N. Current issues in postoperative pain management. Eur J Anaesthesiol. 2016 Mar;33(3):160-71. doi: 10.1097/EJA.0000000000000366. PMID 26509324
- [Result] Weinbroum AA. Superiority of postoperative epidural over intravenous patient-controlled analgesia in orthopedic oncologic patients. Surgery. 2005 Nov;138(5):869-76. doi: 10.1016/j.surg.2005.05.004. PMID 16291387